CLINICAL TRIAL: NCT01449058
Title: A Phase Ib Open-label, Multi-center, Dose Escalation and Expansion Study of Orally Administered MEK162 Plus BYL719 in Adult Patients With Selected Advanced Solid Tumors
Brief Title: A Phase Ib Study of MEK162 Plus BYL719 in Adult Patients With Selected Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMEK162X2109; 2011-002578-21 (EudraCT Number)
Record Dates: First submitted 2011-10-06; First posted 2011-10-07 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Advanced and Selected Solid Tumors; AML; High Risk and Very High Risk MDS
Keywords: Advanced solid tumor,; AML; high risk and very high risk MDS; dose escalation,; RAS/BRAF mutation,; PI3K inhibitor,; MEK inhibitor,; BYL719,; MEK162
MeSH Terms: interventions — Alpelisib; binimetinib

ARMS (1):
- BYL719 + MEK162 (Experimental): BYL719 plus MEK162. Dose escalation with a starting dose for the first cohort of 200mg QD BYL719 and 30mg BID MEK162
  Interventions: Drug: BYL719; Drug: MEK162

INTERVENTIONS:
Drug: BYL719 — taken orally
Drug: MEK162 — taken orally

SUMMARY:
This is a multi-center, open-label, dose-finding, phase Ib study to estimate the maximum tolerated dose(s) (MTD(s)) and/or recommended dose(s) for expansion (RDE(s)) for the orally administered combination of BYL719 and MEK162. This combination will be explored in adult patients with advanced CRC, esophageal cancer, pancreatic cancer, NSCLC, ovarian cancer, or other advanced solid tumors and in adult patients with AML or high risk and very high risk MDS, with documented RAS or BRAF mutations. Dose escalation will be guided by a Bayesian logistic regression model with overdose control. At MTD or RDE, four expansion arms will be opened in order to further assess the safety and preliminary activity of the combination of BYL719 and MEK162 in specific patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed, advanced solid tumors, AML or high risk and very high risk MDS
* Measurable disease as determined by RECIST 1.1

Exclusion Criteria:

* Primary CNS tumor or CNS tumor involvement
* Diabetes mellitus
* Unacceptable ocular/retinal conditions
* Clinically significant cardiac disease or impaired cardiac function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2012-03; Primary Completion 2016-08-31 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLT) | during the first cycle (28 days) of treatment with BYL719 and MEK162
  Toxicity will be assessed using the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), version 4.0 unless otherwise specified. A DLT is defined as an adverse event or abnormal laboratory value assessed as at least possibly related to the study medication, occurs ≤ 28 days following the first dose of BYL719 and MEK162 (Cycle 1), and meets any of the protocol-specified DLT criteria.

SECONDARY OUTCOMES:
Number of participants with adverse events and serious adverse events | Assessed from Cycle 1 Day 1 until treatment discontinuation
  All AEs and SAEs will be collected in accordance with the protocol and assessed for relatedness to study drug combination.
Overall response rate | Assessed every 8 weeks until disease progression
  Overall response rate (ORR) is the proportion of patients with a best overall response of Complete Response (CR) or Partial Response (PR).
Time to progression | Assessed every 8 weeks until disease progression
  Time to progression (TTP) is the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to underlying cancer. If a patient has not had an event, time to progression is censored at the date of last adequate tumor assessment.
Progression free survival | Assessed every 8 weeks until disease progression
  Progression-free survival (PFS) is the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient has not had an event, progression-free survival is censored at the date of last adequate tumor assessment.
Time versus plasma concentration profiles of BYL719 and MEK162 | Assessed during the first cycle of treatment
  Blood concentrations of MEK162 and its metabolite (AR00426032) and BYL719 will be assessed during the first cycle of treatment.
Correlation of baseline mutation or amplification status (PIK3CA, KRAS, NRAS and BRAF) and clinical anti-tumor activity outcome | Assessed at Baseline (pre-treatment)
  Collect baseline genetic mutation/alteration status to investigate the potential relationship to anti-tumor activity.
Clinical benefit rate | Assessed every 4 weeks for 3 months and every 3 months for 6 months followed by every 6 months thereafter until disease progression
  The clinical benefit rate is defined as the proportion of patients with complete remission, complete remission with incomplete blood count recovery, partial remission, minor response or stable disease for > 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Array BioPharma, Study Director — 303-381-6604
Locations (15):
- United States (8):
  - University of California San Diego - Moores Cancer Center Dept Onc, La Jolla, California
  - H. Lee Moffitt Cancer Center & Research Institute H. Lee Moffitt SC, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Massachusetts General Hospital CCPO, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center Onc. Dept, New York, New York
  - Montefiore Medical Center SC, The Bronx, New York
  - University of Texas/MD Anderson Cancer Center Dept. of Onc., Houston, Texas
  - University of Utah / Huntsman Cancer Institute Huntsman (3), Salt Lake City, Utah
- Array BioPharma Investigative Site, Parkville, Victoria, Australia
- Array BioPharma Investigative Site, Villejuif, France
- Italy (2):
  - Array BioPharma Investigative Site, Milan, MI
  - Array BioPharma Investigative Site, Roma, RM
- Array BioPharma Investigative Site, Barcelona, Catalonia, Spain
- Array BioPharma Investigative Site, Bellinzona, Switzerland
- Array BioPharma Investigative Site, Sutton, United Kingdom